CLINICAL TRIAL: NCT05951231
Title: Liver Transplantation After ex Vivo Liver Perfusion - The EVOLVE Study
Brief Title: Liver Transplantation After ex Vivo Liver Perfusion
Acronym: EVOLVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Søren Erik Pischke, Principal investigator, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 598448
Record Dates: First submitted 2023-04-04; First posted 2023-07-18 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Liver Transplant; Complications; Transplant; Failure, Liver; Transplant Dysfunction; Transplant; Complication, Rejection; Transplant; Liver Metastases; Liver Cancer
Keywords: Liver; Transplantation; Perfusion; Dual-end-ischemic Hypothermic Oxygenated Perfusion; Normothermic Machine Perfusion; Controlled Oxygenated Rewarming; Microdialysis
MeSH Terms: conditions — Rejection, Psychology; Liver Neoplasms | interventions — Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Single center, prospective, open, observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver transplanted patient (Active Comparator): Patients who are transplanted with an ECD liver after pretreatment with a liver perfusion machine
  Interventions: Procedure: Liver transplantation
- Non-liver transplanted patient (No Intervention): Patients who are not offered a liver transplantation during the inclusion period

INTERVENTIONS:
Procedure: Liver transplantation — Patients who receive an ECD liver after an ex-vivo liver perfusion where the liver has been tested for function and approved according to international functional criteria (Groeningen criteria)
  Arms: Liver transplanted patient

SUMMARY:
Today, it is difficult to predict liver function after transplantation and therefore livers where poor function is assumed (marginal livers) become discarded. The study aim is to increase the number of available donor livers, especially for liver cancer patients, by pre-treating and testing marginal ones (extended criteria donor (ECD) livers) liver on a liver perfusion machine. A liver perfusion machine can simulate liver transplantation and enables functional/quality testing before transplantation. The machine will hopefully also make marginal livers more functional by reducing ischemia- & reperfusion injury. A marginal donor liver is perfused ex situ with oxygenated blood from a blood donor on a machine. The liver can be tested here for function using internationally recognized criteria. At the same time, the investigators will carry out analyzes with microdialysis which can give a better picture of organ function and damage. Additionally, various samples of the liver and perfusate will be collected. Liver that achieves criteria for transplantation will be offered to the recipient.

DETAILED DESCRIPTION:
The study is a single-center, prospective, open-label cohort study designed to determine the efficacy of liver perfusion of marginal ECD livers on a perfusion machine before liver transplantation. Donor livers will be preserved with standard cooling followed by three perfusion modes (Dual hypothermic oxygenated machine perfusion (DHOPE) / Controlled oxygenated rewarming (COR) / Normothermic machine perfusion (NMP)), a method used internationally to pre-treating marginal livers before liver transplantation and which able testing of function and quality before a transplantation is performed. Only livers that fulfill international criteria (Groningen criteria) will be approved for Ltx. In this study microdialysis will be used to monitoring the liver during machine perfusion and up to 14 days in the postoperative course to monitor the function of the liver. The hypothesis is that microdialysis will provide a better prediction of liver function than the existing Groeningen criteria. The investigators expect that most included patients, who receive ECD livers perfused on a machine, will receive a postoperative well-functioning liver graft which entails a significant survival benefit. The study is designed as a cohort study because included patients have a very poor prognosis (median overall survival of approx. 6 months) and others treatment options are lacking. The primary objective is to establish definitive, objective criteria for pre-transplant liver function by defining a threshold value for microdialysis parameters (especially lactate) between donor livers that will restore function and those that will not during ex vivo machine perfusion in ECD livers, which are superior to established criteria (Groeningen and Viability testing and transplantation of marginal livers (VITTAL) criteria)). The primary endpoint is microdialysis lactate level between donor livers after 4 hours of normothermic machine perfusion in ECD livers.

The follow-up period is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* ≥ 18 years
* Indication for liver transplantation (one criteria must be met):
* Colorectal cancer patients who have received 1st and 2nd line chemotherapy where the treatment has been stopped due to progression or toxicity and the patient is not eligible for SECA-2 (Survival Following Liver Transplantation for Patients With Nonresectable Liver-only Colorectal Metastases) study.
* Hepatocellular carcinoma patients who are not suitable for standard liver transplantation, liver resection or local treatment (Transarterial Chemoembolisation or Selective internal radiotherapy). The patients must have progression or intolerance (toxicity) for immune checkpoint inhibitors or 1st line treatment.
* Cholangiocarcinoma patients who have progression or intolerance to first-line chemotherapy.
* Benign liver disease with urgent need for transplantation within months, but no regular graft is available.
* Life expectancy ≤ 6 months
* Willing, able and expected cooperation to attend follow-up examinations
* Patients who have a need for liver transplantation but cannot participate in other transplant studies or participation in another clinical trial with randomization to liver transplantation.

For malignant disease the following criteria must be met:

* Good performance status assessed at the discretion of the treating physician.
* ECOG (Eastern Cooperative Oncology Group) 0 or 1
* Satisfactory blood tests

  * Hemoglobin >8 g/dl
  * Neutrophiles >1.0 (after any Granulocyte colony-stimulating factor)
  * Platelets >75
  * Bilirubin <1.5 x upper normal level
  * ASAT (Aspartate aminotransferase), ALAT (alanine aminotransferase) <5 x upper normal level
  * Albumin above lower normal level.

Exclusion Criteria:

* Already listed for ordinary Ltx with expectance of getting offered a regular liver graft within a reasonable time-frame.
* Patients included in the control arm of the SECA-3 study or the Excalibur studies except for the Ltx arm of the Excalibur I study.
* Mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Lactate level in microdialysate from hilar plate after normothermic machine perfusion - 4 hours | 4 hours
  Lactate level in microdialysate from hilar plate after normothermic machine perfusion in extended criteria donors livers.

SECONDARY OUTCOMES:
Lactate level in microdialysate from liver tissue after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Microdialysis lactate level in donor liver tissue after 2.5 hours of normothermic machine perfusion in extended criteria donors livers.
Lactate level in microdialysate from liver tissue after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Microdialysis lactate level in donor liver tissue after 2 hours of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Pyruvate level in microdialysate from liver tissue after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Microdialysis pyruvate level in donor liver tissue after 2 hours of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Glycerol level in microdialysate from liver tissue after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Microdialysis glycerol level in donor liver tissue after 2 hours of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Glucose level in microdialysate from liver tissue after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Microdialysis glucose level in donor liver tissue after 2 hours of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Lactate level in microdialysate from liver tissue after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Microdialysis lactate level in donor livers tissue after 1 hour of controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Glycerol level in microdialysate from liver tissue after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Microdialysis glycerol level in donor livers tissue after 1 hour of controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Glucose level in microdialysate from liver tissue after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Microdialysis glucose level in donor livers tissue after 1 hour of controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Pyruvate level in microdialysate from liver tissue after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Microdialysis pyruvate level in donor livers tissue after 1 hour of controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Glucose level in microdialysate from liver tissue after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Microdialysis glucose level in donor liver tissue after 2.5 hours of normothermic machine perfusion in extended criteria donors livers.
Glucose level in microdialysate from liver tissue after normothermic machine perfusion - 4 hours | 4 hours
  Microdialysis glucose level in donor liver tissue after 4 hours of normothermic machine perfusion in extended criteria donors livers.
Pyruvate level in microdialysate from liver tissue after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Microdialysis pyruvate level in donor liver tissue after 2.5 hours of normothermic machine perfusion in extended criteria donors livers.
Pyruvate level in microdialysate from liver tissue after normothermic machine perfusion - 4 hours | 4 hours
  Microdialysis pyruvate level in donor liver tissue after 4 hours of normothermic machine perfusion in extended criteria donors livers.
Glycerol level in microdialysate from liver tissue after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Microdialysis glycerol level in donor liver tissue after 2.5 hours of normothermic machine perfusion in extended criteria donors livers.
Glycerol level in microdialysate from liver tissue after normothermic machine perfusion - 4 hours | 4 hours
  Microdialysis glycerol level in donor liver tissue after 4 hours of normothermic machine perfusion in extended criteria donors livers.
Lactate level in microdialysate from bile after normothermic machine perfusion - 4 hours | 4 hours
  Microdialysis lactate level from bile after normothermic machine perfusion - 4 hours in extended criteria donors livers.
Lactate level in microdialysate from bile after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Microdialysis lactate level from bile after normothermic machine perfusion - 2.5 hours in extended criteria donors livers.
Glucose level in microdialysate from bile after normothermic machine perfusion - 4 hours | 4 hours
  Microdialysis glucose levels from bile after normothermic machine perfusion - 4 hours in extended criteria donors livers.
Glucose level in microdialysate from bile after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Microdialysis glucose levels from bile after normothermic machine perfusion - 2.5 hours in extended criteria donors livers.
Pyruvate level in microdialysate from bile after normothermic machine perfusion - 4 hours | 4 hours
  Microdialysis pyruvate levels from bile after normothermic machine perfusion - 4 hours in extended criteria donors livers.
Pyruvate level in microdialysate from bile after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Microdialysis pyruvate levels from bile after normothermic machine perfusion - 2.5 hours in extended criteria donors livers.
Glycerol level in microdialysate from bile after normothermic machine perfusion - 4 hours | 4 hours
  Glycerol levels from bile after normothermic machine perfusion - 4 hours in extended criteria donors livers.
Glycerol level in microdialysate from bile after normothermic machine perfusion - 2.5 hours | 2.5 hours
  Glycerol levels from bile after normothermic machine perfusion - 2.5 hours in extended criteria donors livers.
Glycerol level in microdialysate from bile after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Glycerol levels from bile after controlled oxygenated rewarming machine perfusion - 1 hour - in extended criteria donors livers.
Glucose level in microdialysate from bile after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Glucose levels from bile after controlled oxygenated rewarming machine perfusion - 1 hour - in extended criteria donors livers.
Lactate level in microdialysate from bile after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Lactate levels from bile after controlled oxygenated rewarming machine perfusion - 1 hour - in extended criteria donors livers.
Pyruvate level in microdialysate from bile after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Pyruvate levels from bile after controlled oxygenated rewarming machine perfusion - 1 hour - in extended criteria donors livers.
Pyruvate level in microdialysate from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Pyruvate levels from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours - in extended criteria donors livers.
Glycerol level in microdialysate from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Glycerol levels from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours - in extended criteria donors livers.
Lactate level in microdialysate from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Lactate levels from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours - in extended criteria donors livers.
Glucose level in microdialysate from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Glucose levels from bile after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours - in extended criteria donors livers.
Bile gases pH - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas pH - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases pH - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas pH - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Lactate - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas Lactate - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Lactate - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas Lactate - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Glucose - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas Glucose - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Glucose - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas Glucose - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Oxygen (O2) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas O2 - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases O2 - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas O2 - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases carbon dioxide (CO2) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas CO2 - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases CO2 - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas CO2 - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases bicarbonate (HCO3) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas HCO3 - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases HCO3 - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas HCO3 - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases base excess (BE) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas BE - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Ischemia/reperfusion injury - 4 hours after normothermic machine perfusion | 4 hours
  Ischemia/reperfusion injury in liver biopsies, graded according to Ali JM et al, Liver transplant 2015; nil, mild, moderate, and severe. - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Ischemia/reperfusion damage - 4 hours after normothermic machine perfusion | 4 hours
  Ischemia/reperfusion damage in liver biopsies, graded according to Suzuki score (Tian Y et al, Stem Cell Research & Therapy, 2016); score 0, 1, 2, 3, (0=none, 4= severe) - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Ischemia/reperfusion injury - after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 4 hours
  Ischemia/reperfusion injury in liver biopsies, graded according to Tian Y et al et al, Liver transplant 2015; nil, mild, moderate, and severe. - after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Ischemia/reperfusion damage - after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 4 hours
  Ischemia/reperfusion damage in liver biopsies, graded according to Suzuki score (Tian Y et al, Stem Cell Research & Therapy, 2016); score 0, 1, 2, 3, (0=none, 4= severe) - after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Ischemia/reperfusion injury - before machine perfusion | 1 minute
  Ischemia/reperfusion injury in liver biopsies, graded according to Ali JM et al, Liver transplant 2015; nil, mild, moderate, and severe. - before machine perfusion in extended criteria donors livers
Ischemia/reperfusion damage - before machine perfusion | 1 minute
  Ischemia/reperfusion damage in liver biopsies, graded according to Suzuki score (Tian Y et al, Stem Cell Research & Therapy, 2016); score 0, 1, 2, 3, (0=none, 4= severe) - before machine perfusion in extended criteria donors livers
Ischemia/reperfusion injury - after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Ischemia/reperfusion injury in liver biopsies, graded according to Ali JM et al, Liver transplant 2015; nil, mild, moderate, and severe - after controlled oxygenated rewarming machine perfusion - 1 hour in extended criteria donors livers
Ischemia/reperfusion damage - after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Ischemia/reperfusion damage in liver biopsies, graded according to Suzuki score (Tian Y et al, Stem Cell Research & Therapy, 2016); score 0, 1, 2, 3, (0=none, 4= severe) - after controlled oxygenated rewarming machine perfusion - 1 hour in extended criteria donors livers
Ischemia/reperfusion injury - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Ischemia/reperfusion injury in liver biopsies, graded according to Ali JM et al, Liver transplant 2015; nil, mild, moderate, and severe. - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Ischemia/reperfusion damage - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Ischemia/reperfusion damage in liver biopsies, graded according to Suzuki score (Tian Y et al, Stem Cell Research & Therapy, 2016); score 0, 1, 2, 3, (0=none, 4= severe) - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases BE - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas BE - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases oxygen saturation (SO2) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas SO2- 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases SO2 - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas SO2- 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases hemoglobin (Hb)- 4 hours after normothermic machine perfusion | 4 hours
  Bile gas Hb - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Hb - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas Hb - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases sodium (Na) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas Na - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Na - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas Na - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases potassium (K) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas K - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases K - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas K - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Calcium (Ca) - 4 hours after normothermic machine perfusion | 4 hours
  Bile gas Ca - 4 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gases Ca - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Bile gas Ca - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Markers of injury, inflammation - 2.5 hours after normothermic machine perfusion | 2.5 hours
  Markers of injury, inflammation - 2.5 hours after normothermic machine perfusion in extended criteria donors livers.
Bile gas lactate 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas lactate 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Markers of injury, inflammation 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Markers of injury, inflammation 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas Glucose 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas Glucose 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas pH 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas pH 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas O2 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas O2 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas CO2 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas CO2 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas HCO3 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas HCO3 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas SO2 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas SO2 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas Hemoglobin 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas Hemoglobin 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas Na 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas Na 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas K 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas K 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas Ca 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas Ca 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Bile gas BE 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion | 2 hours
  Bile gas BE 2 hours after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Markers of injury, inflammation 1 hour after controlled oxygenated rewarming machine perfusion | 1 hour
  Markers of injury, inflammation 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas lactate 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas lactate 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas Glucose 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas Glucose 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas pH 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas pH 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Markers of injury, inflammation 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Markers of injury, inflammation 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas O2 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas O2 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas CO2 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas CO2 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas HCO3 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas HCO3 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas BE 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas BE 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas SO2 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas SO2 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas hemoglobin 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas hemoglobin 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas Na 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas Na 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas K 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas K 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Bile gas Ca 1 hour after controlled oxygenated rewarming machine perfusion | 1 hours
  Bile gas Ca 1 hour after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Perfusate gas Ca - during machine perfusion | 24 hours
  Perfusate gas Ca during machine perfusion in extended criteria donors livers.
Perfusate gas pH - during machine perfusion | 24 hours
  Perfusate gas pH during machine perfusion in extended criteria donors livers.
Perfusate gas SO2 - during machine perfusion | 24 hours
  Perfusate gas SO2 during machine perfusion in extended criteria donors livers.
Perfusate gas O2 - during machine perfusion | 24 hours
  Perfusate gas O2 during machine perfusion in extended criteria donors livers.
Perfusate gas CO2 - during machine perfusion | 24 hours
  Perfusate gas CO2 during machine perfusion in extended criteria donors livers.
Perfusate gas K - during machine perfusion | 24 hours
  Perfusate gas K during machine perfusion in extended criteria donors livers.
Perfusate gas Na - during machine perfusion | 24 hours
  Perfusate gas Na during machine perfusion in extended criteria donors livers.
Perfusate gas BE - during machine perfusion | 24 hours
  Perfusate gas BE during machine perfusion in extended criteria donors livers.
Perfusate gas HCO3 - during machine perfusion | 24 hours
  Perfusate gas HCO3 during machine perfusion in extended criteria donors livers.
Perfusate gas hemoglobin - during machine perfusion | 24 hours
  Perfusate gas hemoglobin during machine perfusion in extended criteria donors livers.
Perfusate gas lactate - during machine perfusion | 24 hours
  Perfusate gas lactate during machine perfusion in extended criteria donors livers.
Perfusate gas glucose - during machine perfusion | 24 hours
  Perfusate gas glucose during machine perfusion in extended criteria donors livers.
Postoperative complications | 12 months
  According to Clavien Dindo Classification
Length of stay | 4 months
  Length of initial ICU and initial hospital stay is determined in days of admission following liver transplantation.
Machine flow during controlled oxygenated rewarming | 1 hour
  Machine flow (millilitre/hour)
Machine flow during Dual-end-ischemic Hypothermic Oxygenated Perfusion | 1 hour
  Machine flow (millilitre/hour)
Machine pressure during controlled oxygenated rewarming | 1 hour
  Machine pressure ((millimetre Hg))
Machine pressure during Dual-end-ischemic Hypothermic Oxygenated Perfusion | 1 hour
  Machine pressure ((millimetre Hg))
Machine Fraction of oxygen during controlled oxygenated rewarming | 1 hour
  Machine fraction of oxygen (%)
Machine Fraction of oxygen Dual-end-ischemic Hypothermic Oxygenated Perfusion | 1 hour
  Machine fraction of oxygen (%)
Machine Resistance during controlled oxygenated rewarming | 1 hour
  Machine Resistance (millilitre/minute/millimetre Hg)
Machine Resistance during Dual-end-ischemic Hypothermic Oxygenated Perfusion | 1 hour
  Machine Resistance (millilitre/minute/millimetre Hg)
Machine flow during Dual-end-ischemic Hypothermic Oxygenated Perfusion | 2 hours
  Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion flow (millilitre/hour)
Machine flow during normothermic machine perfusion | 4 hours
  Machine flow during normothermic machine perfusion (millilitre/hour)
Machine flow during normothermic machine perfusion | 2.5 hours
  Machine flow during normothermic machine perfusion (millilitre/hour)
Machine pressure during normothermic machine perfusion | 4 hours
  Machine pressure (millimetre Hg)
Machine pressure during normothermic machine perfusion | 2.5 hours
  Machine pressure (millimetre Hg)
Machine Fraction of oxygen during normothermic machine perfusion | 4 hours
  Machine fraction of oxygen (%)
Machine Fraction of oxygen during normothermic machine perfusion | 2.5 hours
  Machine fraction of oxygen (%)
Machine Resistance during normothermic machine perfusion | 4 hours
  Machine Resistance (millilitre/minute/millimetre Hg)
Machine Resistance during normothermic machine perfusion | 2.5 hours
  Machine Resistance (millilitre/minute/millimetre Hg)
Total preservation time | 48 hours
  Total preservation time (machine perfusion time)
Alanine amino transferase in perfusate during machine perfusion | 24 hours
  Alanine amino transferase in perfusate during machine perfusion (U/Litre)
Aspartate amino transferase in perfusate during machine perfusion | 24 hours
  Aspartate amino transferase in perfusate during machine perfusion (U/Litre)
Alkaline phosphatase in perfusate during machine perfusion | 24 hours
  Aspartate amino transferase in perfusate during machine perfusion (U/Litre)
Gamma-glutamyl transferase in perfusate during machine perfusion | 24 hours
  Gamma-glutamyl transferase in perfusate during machine perfusion (U/Litre)
Urea in perfusate during machine perfusion | 24 hours
  Urea in perfusate during machine perfusion (millimol/Litre)
Bilirubin in perfusate during machine perfusion | 24 hours
  Bilirubin in perfusate during machine perfusion (micromol/Litre)
Not yet decided types of cytokines/interleukins, endothelium markers, miRNA's in perfusate during machine perfusion | 24 hours
  Different cytokines/interleukins, endothelium markers, miRNA's in perfusate during machine perfusion
Not yet decided types of cytokines/interleukins, endothelium markers, miRNA's in liver tissue during machine perfusion | 24 hours
  Different cytokines/interleukins, endothelium markers, miRNA's in liver tissue during machine perfusion
Not yet decided types of cytokines/interleukins, endothelium markers, miRNA's in bile during machine perfusion | 24 hours
  Different cytokines/interleukins, endothelium markers, miRNA's in bile during machine perfusion
Histopathology - liver tissue. Mitochondrial function | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for mitochondrial function.
Histopathology - bile duct. Mitochondrial function | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for mitochondrial function.
Histopathology - liver tissue. Perfusion/reperfusion injury | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for perfusion/reperfusion injury
Histopathology - bile duct. Perfusion/reperfusion injury | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for perfusion/reperfusion injury
Histopathology - liver tissue. Cell death | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for cell death
Histopathology - bile duct. Cell death | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for cell death
Histopathology - liver tissue. Inflammation | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for inflammation
Histopathology - bile duct. Inflammation | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for inflammation
Histopathology - liver tissue. Metabolomics | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for metabolomics
Histopathology - bileduct. Metabolomics | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for metabolomics
Histopathology - liver tissue. Lipidomics | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for lipidomics
Histopathology - bile duct. Lipidomics | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for lipidomics
Histopathology - liver tissue. RNA sequencing | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for RNA sequencing
Histopathology - bile duct. RNA sequencing | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for RNA sequencing
Histopathology - liver tissue. Endothelium properties | During machine perfusion - 24 hours
  Histological analysis of parenchymal biopsies which are assessed for endothelium properties
Histopathology - bile duct. Endothelium properties | During machine perfusion - 24 hours
  Histological analysis of bile duct biopsies which are assessed for endothelium properties
International normalized ratio on postoperative day 7 | 7 postoperative day
  Blood sample from recipient: International normalized ratio on postoperative day 7
Alanine amino transferase postoperative day 0 | Postoperative day 0
  Alanine amino transferase postoperative day 0 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative day 0 | Postoperative day 0
  Aspartate amino transferase postoperative day 0 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 0 | Postoperative day 0
  Alkaline phosphatase postoperative day 0 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 0 | Postoperative day 0
  Gamma-glutamyl transferase postoperative day 0 in the donated recipients (U/Litre)
Urea postoperative day 0 | Postoperative day 0
  Urea postoperative day 0 in the donated recipients (millimol/Litre)
Bilirubin postoperative day 0 | Postoperative day 0
  Bilirubin postoperative day 0 in the donated recipients (micromol/Litre)
Bilirubin postoperative day 1 | Postoperative day 1
  Bilirubin postoperative day 1 in the donated recipients (micromol/Litre)
Bilirubin postoperative day 2 | Postoperative day 2
  Bilirubin postoperative day 2 in the donated recipients (micromol/Litre)
Bilirubin postoperative day 3 | Postoperative day 3
  Bilirubin postoperative day 3 in the donated recipients (micromol/Litre)
Bilirubin postoperative day 4 | Postoperative day 4
  Bilirubin postoperative day 4 in the donated recipients (micromol/Litre)
Bilirubin postoperative day 5 | Postoperative day 5
  Bilirubin postoperative day 5 in the donated recipients (micromol/Litre)
Bilirubin postoperative day 6 | Postoperative day 6
  Bilirubin postoperative day 6 in the donated recipients (micromol/Litre)
Bilirubin postoperative day 7 | Postoperative day 7
  Bilirubin postoperative day 7 in the donated recipients (micromol/Litre)
Urea postoperative day 1 | Postoperative day 1
  Urea postoperative day 1 in the donated recipients (millimol/Litre)
Urea postoperative day 2 | Postoperative day 2
  Urea postoperative day 2 in the donated recipients (millimol/Litre)
Urea postoperative day 3 | Postoperative day 3
  Urea postoperative day 3 in the donated recipients (millimol/Litre)
Urea postoperative day 4 | Postoperative day 4
  Urea postoperative day 4 in the donated recipients (millimol/Litre)
Urea postoperative day 5 | Postoperative day 5
  Urea postoperative day 5 in the donated recipients (millimol/Litre)
Urea postoperative day 6 | Postoperative day 6
  Urea postoperative day 6 in the donated recipients (millimol/Litre)
Urea postoperative day 7 | Postoperative day 7
  Urea postoperative day 7 in the donated recipients (millimol/Litre)
Aspartate amino transferase postoperative day 1 | Postoperative day 1
  Aspartate amino transferase postoperative day 1 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 1 | Postoperative day 1
  Alkaline phosphatase postoperative day 1 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 1 | Postoperative day 1
  Gamma-glutamyl transferase postoperative day 1 in the donated recipients (U/Litre)
Alanine amino transferase postoperative day 2 | Postoperative day 2
  Alanine amino transferase postoperative day 2 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative day 2 | Postoperative day 2
  Aspartate amino transferase postoperative day 2 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 2 | Postoperative day 2
  Alkaline phosphatase postoperative day 2 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 2 | Postoperative day 2
  Gamma-glutamyl transferase postoperative day 2 in the donated recipients (U/Litre)
Alanine amino transferase postoperative day 3 | Postoperative day 3
  Alanine amino transferase postoperative day 3 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative day 3 | Postoperative day 3
  Aspartate amino transferase postoperative day 3 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 3 | Postoperative day 3
  Alkaline phosphatase postoperative day 3 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 3 | Postoperative day 3
  Gamma-glutamyl transferase postoperative day 3 in the donated recipients (U/Litre)
Alanine amino transferase postoperative day 4 | Postoperative day 4
  Alanine amino transferase postoperative day 4 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative day 4 | Postoperative day 4
  Aspartate amino transferase postoperative day 4 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 4 | Postoperative day 4
  Alkaline phosphatase postoperative day 4 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 4 | Postoperative day 4
  Gamma-glutamyl transferase postoperative day 4 in the donated recipients (U/Litre)
Alanine amino transferase postoperative day 5 | Postoperative day 5
  Alanine amino transferase postoperative day 5 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative day 5 | Postoperative day 5
  Aspartate amino transferase postoperative day 5 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 5 | Postoperative day 5
  Alkaline phosphatase postoperative day 5 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 5 | Postoperative day 5
  Gamma-glutamyl transferase postoperative day 5 in the donated recipients (U/Litre)
Alanine amino transferase postoperative day 6 | Postoperative day 6
  Alanine amino transferase postoperative day 6 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative day 6 | Postoperative day 6
  Aspartate amino transferase postoperative day 6 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 6 | Postoperative day 6
  Aspartate amino transferase postoperative day 6 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 6 | Postoperative day 6
  Gamma-glutamyl transferase postoperative day 6 in the donated recipients (U/Litre)
Alanine amino transferase postoperative day 7 | Postoperative day 7
  Alanine amino transferase postoperative day 7 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative day 7 | Postoperative day 7
  Aspartate amino transferase postoperative day 7 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative day 7 | Postoperative day 7
  Alkaline phosphatase postoperative day 7 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative day 7 | Postoperative day 7
  Gamma-glutamyl transferase postoperative day 7 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 1 | 1 month after surgery
  Alanine amino transferase postoperative month 1 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 1 | 1 month after surgery
  Aspartate amino transferase postoperative month 1 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 1 | 1 month after surgery
  Alkaline phosphatase postoperative month 1 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 1 | 1 month after surgery
  Gamma-glutamyl transferase postoperative month 1 in the donated recipients (U/Litre)
Urea postoperative month 1 | 1 month after surgery
  Urea postoperative month 1 in the donated recipients (millimol/Litre)
Bilirubin postoperative month 1 | 1 month after surgery
  Bilirubin postoperative month 1 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 2 | 2 month after surgery
  Bilirubin postoperative month 2 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 3 | 3 month after surgery
  Bilirubin postoperative month 3 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 4 | 4 month after surgery
  Bilirubin postoperative month 4 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 5 | 5 month after surgery
  Bilirubin postoperative month 5 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 6 | 6 month after surgery
  Bilirubin postoperative month 6 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 7 | 7 month after surgery
  Bilirubin postoperative month 7 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 8 | 8 month after surgery
  Bilirubin postoperative month 8 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 9 | 9 month after surgery
  Bilirubin postoperative month 9 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 10 | 10 month after surgery
  Bilirubin postoperative month 10 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 11 | 11 month after surgery
  Bilirubin postoperative month 11 in the donated recipients (micromol/Litre)
Bilirubin postoperative month 12 | 12 month after surgery
  Bilirubin postoperative month 12 in the donated recipients (micromol/Litre)
Urea postoperative month 2 | 2 month after surgery
  Urea postoperative month 2 in the donated recipients (millimol/Litre)
Urea postoperative month 3 | 3 month after surgery
  Urea postoperative month 3 in the donated recipients (millimol/Litre)
Urea postoperative month 4 | 4 month after surgery
  Urea postoperative month 4 in the donated recipients (millimol/Litre)
Urea postoperative month 5 | 5 month after surgery
  Urea postoperative month 5 in the donated recipients (millimol/Litre)
Urea postoperative month 6 | 6 month after surgery
  Urea postoperative month 6 in the donated recipients (millimol/Litre)
Urea postoperative month 7 | 7 month after surgery
  Urea postoperative month 7 in the donated recipients (millimol/Litre)
Urea postoperative month 8 | 8 month after surgery
  Urea postoperative month 8 in the donated recipients (millimol/Litre)
Urea postoperative month 9 | 9 month after surgery
  Urea postoperative month 9 in the donated recipients (millimol/Litre)
Urea postoperative month 10 | 10 month after surgery
  Urea postoperative month 10 in the donated recipients (millimol/Litre)
Urea postoperative month 11 | 11 month after surgery
  Urea postoperative month 11 in the donated recipients (millimol/Litre)
Urea postoperative month 12 | 12 month after surgery
  Urea postoperative month 12 in the donated recipients (millimol/Litre)
Alanine amino transferase postoperative month 2 | 2 month after surgery
  Alanine amino transferase postoperative month 2 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 2 | 2 month after surgery
  Aspartate amino transferase postoperative month 2 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 2 | 2 month after surgery
  Alkaline phosphatase postoperative month 2 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 2 | 2 month after surgery
  Gamma-glutamyl transferase postoperative month 2 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 3 | 3 month after surgery
  Alanine amino transferase postoperative month 3 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 3 | 3 month after surgery
  Aspartate amino transferase postoperative month 3 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 3 | 3 month after surgery
  Alkaline phosphatase postoperative month 3 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 3 | 3 month after surgery
  Gamma-glutamyl transferase postoperative month 3 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 4 | 4 month after surgery
  Alanine amino transferase postoperative month 4 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 4 | 4 month after surgery
  Aspartate amino transferase postoperative month 4 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 4 | 4 month after surgery
  Alkaline phosphatase postoperative month 4 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 4 | 4 month after surgery
  Gamma-glutamyl transferase postoperative month 4 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 5 | 5 month after surgery
  Alanine amino transferase postoperative month 5 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 5 | 5 month after surgery
  Aspartate amino transferase postoperative month 5 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 5 | 5 month after surgery
  Alkaline phosphatase postoperative month 5 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 5 | 5 month after surgery
  Gamma-glutamyl transferase postoperative month 5 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 6 | 6 month after surgery
  Alanine amino transferase postoperative month 6 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 6 | 6 month after surgery
  Aspartate amino transferase postoperative month 6 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 6 | 6 month after surgery
  Alkaline phosphatase postoperative month 6 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 6 | 6 month after surgery
  Gamma-glutamyl transferase postoperative month 6 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 7 | 7 month after surgery
  Alanine amino transferase postoperative month 7 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 7 | 7 month after surgery
  Aspartate amino transferase postoperative month 7 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 7 | 7 month after surgery
  Alkaline phosphatase postoperative month 7 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 7 | 7 month after surgery
  Gamma-glutamyl transferase postoperative month 7 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 8 | 8 month after surgery
  Alanine amino transferase postoperative month 8 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 8 | 8 month after surgery
  Aspartate amino transferase postoperative month 8 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 8 | 8 month after surgery
  Alkaline phosphatase postoperative month 8 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 8 | 8 month after surgery
  Gamma-glutamyl transferase postoperative month 8 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 9 | 9 month after surgery
  Alanine amino transferase postoperative month 9 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 9 | 9 month after surgery
  Aspartate amino transferase postoperative month 9 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 9 | 9 month after surgery
  Alkaline phosphatase postoperative month 9 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 9 | 9 month after surgery
  Gamma-glutamyl transferase postoperative month 9 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 10 | 10 month after surgery
  Alanine amino transferase postoperative month 10 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 10 | 10 month after surgery
  Aspartate amino transferase postoperative month 10 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 10 | 10 month after surgery
  Alkaline phosphatase postoperative month 10 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 10 | 10 month after surgery
  Gamma-glutamyl transferase postoperative month 10 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 11 | 11 month after surgery
  Alanine amino transferase postoperative month 11 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 11 | 11 month after surgery
  Aspartate amino transferase postoperative month 11 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 11 | 11 month after surgery
  Alkaline phosphatase postoperative month 11 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 11 | 11 month after surgery
  Gamma-glutamyl transferase postoperative month 11 in the donated recipients (U/Litre)
Alanine amino transferase postoperative month 12 | 12 month after surgery
  Alanine amino transferase postoperative month 12 in the donated recipients (U/Litre)
Aspartate amino transferase postoperative month 12 | 12 month after surgery
  Aspartate amino transferase postoperative month 12 in the donated recipients (U/Litre)
Alkaline phosphatase postoperative month 12 | 12 month after surgery
  Alkaline phosphatase postoperative month 12 in the donated recipients (U/Litre)
Gamma-glutamyl transferase postoperative month 12 | 12 month after surgery
  Gamma-glutamyl transferase postoperative month 12 in the donated recipients (U/Litre)
Postoperative microdialysis levels of lactate | 14 days
  Postoperative microdialysis levels of lactate in transplanted livers the first 14 postoperative days
Postoperative microdialysis levels of pyruvate | 14 days
  Postoperative microdialysis levels of pyruvate in transplanted livers the first 14 postoperative days
Postoperative microdialysis levels of glycerol | 14 days
  Postoperative microdialysis levels of glycerol in transplanted livers the first 14 postoperative days
Postoperative microdialysis levels of glucose | 14 days
  Postoperative microdialysis levels of glucose in transplanted livers the first 14 postoperative days
Systolic blood pressure | From 5 min before reperfusion, up to 20 minutes after reperfusion
  Systolic blood pressure (millimeter Hg)
Diastolic blood pressure | From 5 min before reperfusion, up to 20 minutes after reperfusion
  Diastolic blood pressure (millimeter Hg)
Heart rate | From 5 min before reperfusion, up to 20 minutes after reperfusion
  Heart rate (Beats/minute)
Vasopressor dosage | From 5 min before reperfusion, up to 20 minutes after reperfusion
  Vasopressor dosage (microgram/kilogram/minutes)
Patient survival | Through study completion, an average of 12 months
  Patient survival (days)
Graft survival | Through study completion, an average of 12 months
  Graft (censored and uncensored for patient death) survival (days)
Number of deaths | 7 days after transplantation
  Number of deaths first 7 days after transplantation
Number of retransplantation | 7 days after transplantation
  Number of retransplantation first 7 days after transplantation
Incidens of new onset diabetes after transplantation | Through study completion, an average of 12 months
  New onset diabetes after transplantation after transplantation. New onset diabetes after transplantation is defined according to the World Health Organization criteria (Report 2003 S5-20).
Estimated glomerular filtration rate - Renal function | Through study completion, an average of 12 months
  Estimated glomerular filtration rate according to the 4-variable Modification of Diet in Renal Disease equation.
The incidence of symptomatic Non-anastomotic Biliary Strictures | 6 months
  The incidence of symptomatic non-anastomotic biliary strictures
The incidence of asymptomatic Non-anastomotic Biliary Strictures | 6 months
  The incidence of asymptomatic non-anastomotic biliary strictures
The incidence of asymptomatic Non-anastomotic Biliary Strictures | 12 months
  The incidence of asymptomatic non-anastomotic biliary strictures
The incidence of symptomatic Non-anastomotic Biliary Strictures | 12 months
  The incidence of symptomatic non-anastomotic biliary strictures
The severity of Non-anastomotic Biliary Strictures | Through study completion, an average of 12 months
  The severity of Non-anastomotic Biliary Strictures based on a scoring system described by Buis et. al (mild, moderate, or severe)
The location of Non-anastomotic Biliary Strictures | Through study completion, an average of 12 months
  The location of Non-anastomotic Biliary Strictures is assessed by images of the magnetic resonance cholangiopancreatography
The incidence of infections | Through study completion, an average of 12 months
  The incidence of infections leading to administration of antibiotics/antifungal/antiviral treatment
Lactate level in microdialysate from liver tissue - 4 hours | 4 hours
  Microdialysis lactate level in donor liver tissue after 4 hours of normothermic machine perfusion in extended criteria donors livers.
Pyruvate level in microdialysate from hilar plate after normothermic machine perfusion - 4 hours | 4 hours
  Pyruvate level in microdialysate from hilar plate after normothermic machine perfusion in extended criteria donors livers.
Glycerol level in microdialysate from hilar plate after normothermic machine perfusion - 4 hours | 4 hours
  Glycerol level in microdialysate from hilar plate after normothermic machine perfusion in extended criteria donors livers.
Glucose level in microdialysate from hilar plate after normothermic machine perfusion - 4 hours | 4 hours
  Glucose level in microdialysate from hilar plate after normothermic machine perfusion in extended criteria donors livers.
Glycerol level in microdialysate from hilar plate after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Glycerol level in microdialysate from hilar plate after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Lactate level in microdialysate from hilar plate after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion - 2 hours | 2 hours
  Lactate level in microdialysate from hilar plate after Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Glucose level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Glucose level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Pyruvate level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Pyruvate level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Glycerol level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Glycerol level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Lactate level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion - 1 hour | 1 hour
  Lactate level in microdialysate from hilar plate after controlled oxygenated rewarming machine perfusion in extended criteria donors livers.
Glucose level in microdialysate from hilar plate after of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers - 2 hours | 2 hour
  Glucose level in microdialysate from hilar plate after of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.
Pyruvate level in microdialysate from hilar plate after of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers - 2 hours | 2 hour
  Pyruvate level in microdialysate from hilar plate after of Dual-end-ischemic Hypothermic Oxygenated Perfusion machine perfusion in extended criteria donors livers.

OTHER OUTCOMES:
Donor associated variables - age | 1 hour
  Age of the donor (years)
Donor associated variables - liver steatosis | 1 hour
  Assessment of liver steatosis (%)
Donor associated variables - gender | 1 hour
  Gender of donor
Donor associated variables - Body mass index | 1 hour
  Body mass index of donor (kilogram/meter2)
Donor associated variables - weight of the liver | 1 hour
  Weight of the liver (gram)
Ischemia time - warm | 12 hour
  Estimation of warm ischemia time (minutes)
Ischemia time - cold | 12 hour
  Estimation of cold ischemia time (minutes)
Donor associated variables - Donor risk index | 1 hour
  Donor risk index score - Increasing donor risk index is associated with higher discard rates among deceased donor livers procured for transplant. Low value of 1= best prognosis. High value of 40 = worst prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Søren E Pischke, MD, PhD, Principal Investigator — Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No
Due to Norwegian laws individual participant data are not shared